CLINICAL TRIAL: NCT02142881
Title: Treatment of Masked Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404M49925
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Masked Hypertension; Hypertension; Chronic Renal Insufficiency
MeSH Terms: conditions — Masked Hypertension; Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antihypertensive medication intensification (Experimental)
  Interventions: Other: Antihypertensive medication intensification
- Usual care (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Antihypertensive medication intensification — Antihypertensive medications will be adjusted by study staff based on ambulatory and clinic BP results at baseline and 2 months with a target 24hr systolic blood pressure of <130 mmHg.
  Arms: Antihypertensive medication intensification
Other: Usual care — Antihypertensive medications will be adjusted by the participants' providers (usual care).
  Arms: Usual care

SUMMARY:
To date, most observational and all intervention studies have defined hypertension on the basis of clinic blood pressure (BP). Measurement of BP outside the clinic with home or ambulatory BP provides a better estimate of the risk of cardiovascular disease and all-cause mortality. Using clinic and ambulatory BPs, patients can be categorized as normotensive (normal clinic and ambulatory BPs), white-coat hypertension (elevated clinic BP with normal ambulatory BP), masked hypertension (normal clinic BP with elevated ambulatory BP), and sustained hypertension (elevated clinic and ambulatory BP). Approximately one third of patients with chronic kidney disease (CKD) with normal clinic BP have elevated ambulatory BP (masked hypertension). We demonstrated that, among participants from the Chronic Renal Insufficiency Cohort (CRIC) study, low estimated glomerular filtration rate (eGFR) and elevated proteinuria are associated with increased odds of masked hypertension. Additionally, participants with masked hypertension had increased risk for target organ damage as assessed by left ventricular mass and pulse wave velocity. These results in participants with CKD are consistent with prior studies in patients with normal renal function that demonstrated a two-fold increased risk for cardiovascular events in patients with masked hypertension compared to patients with normal clinic and ambulatory BP. Despite this elevated risk for adverse outcomes, patients with masked hypertension have been excluded from hypertension trials because of their normal clinic BP. Therefore, it is unknown whether the reduction in target organ damage and adverse cardiovascular outcomes associated with treatment of hypertension extends to patients with masked hypertension. To address this important gap in knowledge, we are planning a randomized, controlled trial to evaluate whether antihypertensive treatment can modify BP patterns in patients with masked hypertension, that is, convert them to controlled clinic and ambulatory BP. We will also evaluate the effect antihypertensive treatment on target organ damage in patients with masked hypertension. The current study is a pilot randomized controlled trial to evaluate the feasibility of the planned trial and the effect of antihypertensive therapy on clinic and ambulatory BP, proteinuria, and target organ damage in patients with masked hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* 30 < eGFR < 70 ml/min/1.73m2 within 9 months of the screening visit
* Urine albumin to creatinine ratio >100mg/gm OR a urinalysis with ≥30mg/dL albuminuria within 9 months of the screening visit
* Most recent clinic systolic BP >120 and <140 mmHg within 9 months of the screening visit
* Masked hypertension at the screening and baseline visits
* Clinic systolic BP <140 mmHg
* 24hr ambulatory systolic BP > 130 mmHg
* Taking ≤ 2 antihypertensive medications
* No change in antihypertensive medications for the past 6 months

Exclusion Criteria:

* Heart failure
* Lightheaded with standing
* Loss of consciousness in the past 24 months
* Non-English speakers
* History of breast cancer requiring a mastectomy or radiation on the side of the non-dominant arm and unable or refuses to use the dominant arm for ambulatory BP monitoring
* Cardiovascular event or procedure or hospitalization for unstable angina within the last 3 months
* Inability to perform ambulatory BP monitoring due to compliance or other clinical reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with masked hypertension | 4 months
  Percentage of participants with masked hypertension defined as a 24hr ambulatory systolic blood pressure >130 mmHg and a clinic systolic blood pressure <140 mmHg

SECONDARY OUTCOMES:
Change from baseline in urine albumin to creatinine ratio at 4 months | Baseline, 4 months
Change from baseline in pulse wave velocity at 4 months | Baseline, 4 months
Change from baseline in 24hr ambulatory systolic blood pressure at 4 months | Baseline, 4 months

OTHER OUTCOMES:
Percentage of participants with masked hypertension | 2 months
  Percentage of participants with masked hypertension defined as a 24hr ambulatory systolic blood pressure >130 mmHg and a clinic systolic blood pressure <140 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Drawz, MD, MHS, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States